CLINICAL TRIAL: NCT01193504
Title: Randomized, Masked Comparison of Bromfenac and Besifloxacin BID With Either Prednisolone BID or Loteprednol 0.5% BID for Prevention of Retinal Thickening and CME Following Phacoemulsification
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innovative Medical (Industry)
Responsible Party: Dr. William Trattler, The Center for Excellence in Eye care
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 25324
Record Dates: First submitted 2010-08-31; First posted 2010-09-02 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Pseudophakia; Cataract Surgery
Keywords: Prevention of Retinal Thickening and CME Following Phacoemulsification; Pseudophakia following cataract surgery
MeSH Terms: conditions — Pseudophakia | interventions — prednisolone acetate; Loteprednol Etabonate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pred Forte (Active Comparator): Patients scheduled to undergo phacoemulsification will be randomized in a 1:1 schedule to receive Pred Forte BID for 4 weeks postop. All patients will receive Xibrom BID for one month and Besifloxacin BID for 7 to 10 days postop.
  Interventions: Drug: Pred Forte
- Lotemax (Active Comparator): patients scheduled to undergo phacoemulsification will be randomized in a 1:1 schedule to receive Lotemax BID for 4 weeks postop. All patients will receive Xibrom BID for one month and Besifloxacin BID for 7 to 10 days postop.
  Interventions: Drug: Lotemax

INTERVENTIONS:
Drug: Pred Forte — Pred Forte BID for 4 weeks postop
  Arms: Pred Forte
Drug: Lotemax — Lotemax BID for 4 weeks postop.
  Arms: Lotemax

SUMMARY:
The purpose of this study is to determine if Lotemax eye drops are at least as effective as Pred Forte eye drops, which are the standard of care after cataract surgery.

DETAILED DESCRIPTION:
Prednisolone 1%, a topical steroid, is considered standard of care following cataract surgery to reduce inflammation. We aim to determine if Lotemax is at least as effective as Prednisolone. If so, these findings would demonstrate that physicians have other treatment options to consider.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >18 years of age scheduled to undergo cataract surgery
* Patients with systemic diseases will be enrolled only if there are no ocular manifestations of their disease (e.g. diabetics with normal retinal exams)
* Expected visual outcome of BCVA (best corrected visual acuity)> 20/25 postoperatively, as determined by potential visual acuity testing and review of preoperative corneal topography and OCT (optical coherence tomography).
* Ability to provide informed consent, take study medications as directed, and likely to complete all study visits

Exclusion Criteria:

* Known contraindication to any study medication or any of their components
* Required use of ocular medications other than the study medications during the study
* Evidence of macular disease (Epiretinal membrane, Vitreomacular traction syndrome, macular hole) on preoperative OCT (optical coherence tomography)
* Presence of significant dry macular degeneration that may impact postoperative visual results.
* History of retinal vein occlusion or diabetic macular edema, uveitis or any macular disease predisposing them to cystoid macular edema or prolonged intraocular inflammation.
* Posterior capsule rupture, Vitreous loss during surgery or any other complication that in the surgeon's opinion, could reduce potential for targeted visual outcome
* Anticipated need for mechanical iris dilating devices
* Presence of Epithelial Basement Membrane Dystrophy, significant dry eye, significant blepharitis, or any other corneal condition that may impact BCVA (best corrected visual acuity) postoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Prevention Of Retinal Thickening | 1 Year
  * OCT (optical coherence tomography) with macular thickening
  * Incidence of CME ( cystoids macular edema)
  * BCVA (best corrected visual acuity)
  * UCVA (uncorrected visual acuity)
  * Central corneal thickness

CONTACTS AND LOCATIONS:
Overall Officials: William Trattler, MD, Principal Investigator — The Center for Excellence in Eye Care; John Hovanesian, MD, Principal Investigator — Harvard Eye Associates; Bonnie Henderson, MD, Principal Investigator — Ophthalmic Consultants of Boston
Locations (3):
- United States (3):
  - Harvard Eye Associates, Laguna Hills, California
  - The Center For Excellence in Eye care, Miami, Florida
  - Ophthalmic Consultants of Boston, Waltham, Massachusetts